CLINICAL TRIAL: NCT01494285
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, 3-arm, Parallel-group, Ambulatory Safety and Efficacy Study of ARK-E021 Topical Foam of 5% and 10% in Subjects With Mild to Moderate Acne Vulgaris.
Brief Title: Clinical Study to Evaluate Tolerability and Safety of ARK-E021 Foam and to Monitor Clinical Effect in Acne Vulgaris Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M. Arkin 1999 Ltd. (Other)
Collaborators: Vyne Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MA1001
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Topical; Foam
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARK-E021 5% foam (Experimental)
  Interventions: Drug: ARK-E021 5%
- ARK-E021 10% foam (Experimental)
  Interventions: Drug: ARK-E021 10%
- Placebo foam (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ARK-E021 5% — Topically applied once daily at bedtime
  Other Names: Not yet marketed
  Arms: ARK-E021 5% foam
Drug: ARK-E021 10% — Topically applied once daily at bedtime
  Other Names: Not yet marketed
  Arms: ARK-E021 10% foam
Drug: Placebo — Topically applied once daily at bedtime
  Other Names: Not marketed
  Arms: Placebo foam

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, 3-arm, parallel-group, ambulatory safety and efficacy study of ARK-E021 topical foam of 5% and 10% in subjects with mild to moderate acne vulgaris.

DETAILED DESCRIPTION:
This is a phase I/II prospective, multicenter, randomized, double blind, placebo controlled, parallel group, dose range finding clinical study to evaluate the safety, tolerability and preliminary efficacy of ARK-E021 foam for treatment of acne vulgaris.

It is anticipated that the study will be conducted at the listed Medical Centers as well as out-patient clinics at the community.

Approximately 144 male and female subjects with mild to moderate facial acne vulgaris will be enrolled in this study. Following satisfaction of the entry criteria and screening procedures, subjects will be randomized to either 5% or 10% topical foam (ARK-E021) or placebo foam. Subjects will apply the study medication once daily on the face at bedtime for 12 weeks followed by a post-treatment follow up visit 4 weeks after end of treatment. The first dose will be applied in the presence of the study investigator or his assignee. Subsequent applications will be made by the patient.

Safety will be monitored throughout the study duration. Efficacy will be assessed by facial lesion counts and by the investigator global evaluation of acne severity at baseline and at weeks 3, 6, 9, 12 and 16.

ELIGIBILITY:
Main Inclusion Criteria:

* Patient is male or female between the ages of 12 to 40.
* A clinical diagnosis of acne vulgaris with facial involvement.
* Minimum of 15 inflammatory lesions on the face (papules and/ or pustules)but not more than 40.
* Existence of non-inflammatory lesions on the face (opened and/or closed comedones).
* A score of ≥2 (moderate) on the investigator's global assessment scale.
* Use of non oral contraceptives in female of childbearing potential during the study.
* No known medical conditions that, in the Investigator's opinion could interfere with study participation.
* Patient is willing and able to comply with all the requirement of the study protocol.
* Patient is willing and able to give written informed consent prior to participation in the study.

Main Exclusion Criteria:

* Acne conglobata, acne fulminans, secondary acne (chloracne, drug induced acne), or severe acne requiring systemic treatment.
* One or more active nodule/cyst acne on the face (inactive lesions allowed).
* Excessive facial hair (e.g. beards, sideburns, moustaches, etc.) that would interfere with diagnosis or assessment of acne vulgaris.
* Participation in another investigational drug trial within 30 days prior to study entry.
* Concomitant medication:

  * Use of systemic steroids, systemic antibiotics, systemic treatment for acne vulgaris, systemic anti-inflammatory agents within 4 weeks prior to baseline or during the study.
  * Use of topical steroids, topical antibiotics, topical treatment for acne vulgaris, topical anti-inflammatory agents within 2 weeks prior to baseline or during the study.
  * Treatment for acne with isotretinoin or isotretinoin derivatives within 12 months prior to study entry.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 157 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ARK-E021 topical foam in subjects with acne vulgaris. | Baseline through week 16.
  Subject safety will be assessed following treatment using measurements of the following variables:
  * Physical examination.
  * Vital Signs (HR, BP, Body temperature).
  * Adverse events recording.
  * Concomitant medications.
To evaluate the efficacy of ARK-E021 topical foam in subjects with acne vulgaris. | Baseline through week 16.
  Subject efficacy will be assessed following treatment using measurements of the following variables:
  * Lesion count (inflammatory/non inflammatory and total).
  * Investigator global assessment (IGA; grade 0-4).
  * Lesion documentation by photographs (optional).

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - HaEmek Medical Center, Afula
  - Meir Medical Center, Kfar Saba
  - Souraski Medical Center, Tel Aviv